CLINICAL TRIAL: NCT02178020
Title: Prospective, Randomized Study of Highly-cross Linked Polyethylene vs. Compression Molded Polyethylene for Primary Posterior-stabilized Total Knee Arthroplasty
Brief Title: Outcome Study of Highly-cross Linked Polyethylene vs. Standard Polyethylene for Primary Posterior Stabilized (PS) Total Knee
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Chapel Hill Orthopedics Surgery & Sports Medicine (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: 05017.0501399RC05
Record Dates: First submitted 2014-06-23; First posted 2014-06-30 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Knee Arthroplasty; Osteolysis; Radiolucent Lines
MeSH Terms: conditions — Osteolysis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- knee arthroplasty, standard polyethylene: total knee arthroplasty with Standard Compression Molded tibial Polyethylene Liner
  Interventions: Device: knee arthroplasty, standard polyethylene
- knee arthroplasty, Highly Cross-Linked (XLP) polyethylene: knee arthroplasty with Highly Cross-Linked tibial Polyethylene Liner
  Interventions: Device: knee arthroplasty, XLP polyethylene

INTERVENTIONS:
Device: knee arthroplasty, standard polyethylene — total knee replacement follow-up; clinical and radiographic; revision rate
  Other Names: Zimmer
  Groups: knee arthroplasty, standard polyethylene
Device: knee arthroplasty, XLP polyethylene — total knee arthroplasty with highly crosslinked polyethylene tibial liner
  Other Names: Zimmer: Prolong
  Groups: knee arthroplasty, Highly Cross-Linked (XLP) polyethylene

SUMMARY:
Polyethylene wear and osteolysis remain a concern with the use of modular, fixed bearing total knee arthroplasty. A variety of highly cross-linked polyethylenes have been introduced to decrease this problem, but there is little data on the results and complications of this polyethylene in posterior-stabilized knee prosthesis. The investigators asked the following questions: (1) Are there any differences in the clinical and radiographic results when a highly cross-lined polyethylene is compared to a standard liner? (2) What is the frequency of reoperation in these two groups and are there any specific complications related to highly cross-linked polyethylene liners.

DETAILED DESCRIPTION:
This prospective, randomized study will seek to enroll patients undergoing primary total knee arthroplasty. Preoperative evaluation will include a detailed history and physical exam with clinical data collection (SF-36, WOMAC, and Knee Society Scores), a complete description of the procedure, a demonstration of the actual types of implants and tibial inserts, and an outline of the study protocol and informed consent. Intraoperatively, the patient will undergo a total knee arthroplasty utilizing standard operative procedures. Each patient will receive a Zimmer NexGen posterior-stabilized total knee arthroplasty. During the procedure or preoperative visit, the patient will be randomized by sealed envelope to receive either a standard Zimmer UHMWPE tibial insert or a Zimmer highly cross-linked UHMWPE tibial insert. Both surgeon and patient will be blinded to the type of implant used. there will be no variations in surgical technique and hospital management of the patients throughout the course of the study. Postoperatively, the patient will be seen for routine follow-up at six weeks, 6 months, 1 year and yearly thereafter. Radiographs will be obtained at each visit. Clinical data forms will be completed at each visit. At the conclusion of the study radiographs will be assessed for signs of polyethylene wear, osteolysis and component loosening. the preoperative and postoperative knee scores will be calculated for each patient and compared between the patient groups with standard statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* all patients indicated for primary total posterior stabilized knee arthroplasty

Exclusion Criteria:

* patients who refused participation
* patients who did not comprehend the English language to give informed consent
* patients with severe knee deformity thought to require a primary constrained condylar prosthesis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all female and male patients with arthritis of knee that requires total knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-07; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants requiring revision, or with Device Related Serious Adverse Events | Up to 10 years
  reoperation rate; polyethylene fracture/failure rate
Radiographic osteolysis | up to 10 years
  lucent, periarticular lesions , related to polyethylene wear

SECONDARY OUTCOMES:
knee scores | up to 10 years
  Knee Society Pain and Function scores
knee joint effusion | up to 10 years
  knee joint examination

OTHER OUTCOMES:
LEAS (lower extremity activity score) | up to 10 years
  patient completed activity questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Paul F Lachiewicz, MD, Principal Investigator — Chapel Hill Orthopedic Surgery and Sports Medicine
Locations (1):
- Chapel Hill Orthopedic Surgery and Sports Medicine, Chapel Hill, North Carolina, United States